CLINICAL TRIAL: NCT06283927
Title: The RECSUR-study: Resection Versus Best Oncological Treatment for Recurrent Glioblastoma: Study Protocol for An International Multicenter Prospective Cohort Study (ENCRAM 2302)
Brief Title: The RECSUR-study: Resection Versus Best Oncological Treatment for Recurrent Glioblastoma (ENCRAM 2302)
Acronym: RECSUR
Status: Recruiting | Type: Observational
Sponsor: Jasper Gerritsen (Other)
Collaborators: Haaglanden Medical Centre (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital Heidelberg (Other); Technical University of Munich (Other); Insel Gruppe AG, University Hospital Bern (Other); Massachusetts General Hospital (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Jasper Gerritsen, Dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2020-0812-5
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma, IDH-wildtype; Glioblastoma Multiforme of Brain; Glioblastoma Multiforme, Adult; Recurrent Glioblastoma; Astrocytoma, Malignant; Astrocytoma of Brain
Keywords: Glioblastoma; Radiotherapy; Chemotherapy; Re-resection; Resection; Overall survival; Progression-free survival; Neurological morbidity; Safety; Serious Adverse Events; Quality of life
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Temozolomide; Lomustine; Re-Irradiation; Therapies, Investigational; Immunotherapy; Oncolytic Virotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Re-resection: Resection of the recurrent tumor
  Interventions: Procedure: Re-resection
- Best oncological treatment: Best oncological treatment consisting of re-challenge temozolomide, re-irradiation, experimental therapy, or best supportive care
  Interventions: Drug: Temozolomide; Drug: Lomustine; Radiation: Re-irradiation; Procedure: Experimental therapy; Other: Best supportive care

INTERVENTIONS:
Procedure: Re-resection — Resection of the recurrent tumor
  Groups: Re-resection
Drug: Temozolomide — Re-challenge Temozolomide chemotherapy
  Groups: Best oncological treatment
Drug: Lomustine — Second line chemotherapy with Lomustine
  Groups: Best oncological treatment
Radiation: Re-irradiation — Re-irradiation with single dose, fractionated, or hypofractionated radiation of the recurrent tumor
  Groups: Best oncological treatment
Procedure: Experimental therapy — Experimental phase I therapy with oncolytic virotherapy or immunotherapy (this list is not exhaustive)
  Other Names: Immunotherapy; Oncolytic virotherapy
  Groups: Best oncological treatment
Other: Best supportive care — Best supportive care, focused on alleviating symptoms
  Groups: Best oncological treatment

SUMMARY:
Previous evidence has indicated that resection for recurrent glioblastoma might benefit the prognosis of these patients in terms of overall survival. However, the demonstrated safety profile of this approach is contradictory in the literature and the specific benefits in distinct clinical and molecular patient subgroups remains ill-defined. The aim of this study, therefore, is to compare the effects of resection and best oncological treatment for recurrent glioblastoma as a whole and in clinically important subgroups.

This study is an international, multicenter, prospective observational cohort study. Recurrent glioblastoma patients will undergo tumor resection or best oncological treatment at a 1:1 ratio as decided by the tumor board. Primary endpoints are: 1) proportion of patients with NIHSS (National Institute of Health Stroke Scale) deterioration at 6 weeks after surgery and 2) overall survival. Secondary endpoints are: 1) progression-free survival (PFS), 2) NIHSS deterioration at 3 months and 6 months after surgery, 3) health-related quality of life (HRQoL) at 6 weeks, 3 months, and 6 months after surgery, and 4) frequency and severity of Serious Adverse Events (SAEs) in each arm. Estimated total duration of the study is 5 years. Patient inclusion is 4 years, follow-up is 1 year.

The study has been approved by the Medical Ethics Committee (METC Zuid-West Holland/Erasmus Medical Center; MEC-2020-0812). The results will be published in peer-reviewed academic journals and disseminated to patient organisations and media.

DETAILED DESCRIPTION:
This is an international, multicenter, prospective, cohort study. Eligible patients are operated or receive best oncological treatment with a 1:1 ratio with a sequential computer-generated random number as subject ID. Intraoperative mapping techniques and/or surgical adjuncts can be used in both treatment arms to ensure the safety of the resection (to minimize the risk of postoperative deficits).

Study patients undergo tumor re-resection or receive best oncological treatment and will undergo evaluation at presentation (baseline) and during the follow-up period at 6 weeks, 3 months, and 6 months postoperatively. Motor function will be evaluated using the NIHSS (National Institute of Health Stroke Scale) and MRC (Medical Research Council) scale. Language function will be evaluated using a standard neurolinguistic test-battery consisting of the Aphasia Bedside Check (ABC), Shortened Token test, Verbal fluency, Picture description and Object naming. This neurolinguistic test-battery is the result of a consensus between the participating centers. Cognitive function will be assessed using the Montreal Cognitive Assessment (MOCA). Overall patient functioning with be assessed with the Karnofsky Performance Scale (KPS) and the ASA (American Society of Anesthesiologists) physical status classification system for comorbidities. Health-related quality of life (HRQoL) will be assessed with the EQ-5D questionnaire and the EORTC QLQ-C30 and EORTC QLQ-BN20 questionnaires. Overall survival and progression-free survival will be assessed. We expect to complete patient inclusion in 4 years. The estimated duration of the study, including follow-up, will be 5 years.

The primary study objective is to evaluate the safety and efficacy of re-resection versus best oncological treatment (neurological morbidity and overall survival) in recurrent glioblastoma patients as expressed by NIHSS scores and survival data. Secondary study objectives are to study the overall progressive-free survival (PFS), long-term neurological morbidity (3 months and 6 months postoperatively), health-related quality of life (HRQoL), and Serious Adverse Events (SAEs) after resection versus best oncological treatment as expressed by progression on follow up MRI scans based on the RANO criteria24 for tumor progression; NIHSS scores, quality of life questionnaires (EORTC QLQ C30, EORTC QLQ BN20, EQ-5D), and registration of SAEs.

Patients will be recruited for the study from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals of the ENCRAM Research Consortium, located in Europe and the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Tumor recurrence according to the RANO criteria of a previously diagnosed glioblastoma based on the WHO 2021 classification for glioma
3. The tumor is suitable for resection (according to neurosurgeon)
4. Written informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brainstem, or midline
2. Medical reasons precluding MRI (e.g., pacemaker)
3. Inability to give written informed consent
4. Secondary high-grade glioma due to malignant transformation from low-grade glioma
5. Clinical data unavailable for the newly diagnosed setting

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent glioblastoma will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.
Sampling Method: Non-Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years postoperatively
  Time from diagnosis to death from any cause
Neurological morbidity at 6 weeks | 6 weeks postoperatively
  NIHSS deterioration of 1 point or more at 6 weeks after surgery

SECONDARY OUTCOMES:
Neurological morbidity at 3 months | 3 months postoperatively
  NIHSS deterioration of 1 point or more at 3 months after surgery
Neurological morbidity at 6 months | 6 months postoperatively
  NIHSS deterioration of 1 point or more at 6 months after surgery
Progression-free survival | Up to 5 years postoperatively
  Time from diagnosis to disease progression (occurrence of a new tumor lesions with a volume greater than 0.175 cm3, or an increase in residual tumor volume of more than 25%) or death, whichever comes first
Residual tumor volume | Within 72 hours postoperatively
  Residual tumor volume of the contrast-enhancing and non-contrast enhancing part, as assessed by a neuroradiologist on postoperative MRI scan (T1 with contrast and FLAIR sequences) using manual or semi-automatic volumetric analyses (Brainlab Elements iPlan CMF Segmentation, Brainlab AG, Munich, Germany; or similar software)
Quality of life at 6 weeks (EORTC QLQ C30) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 3 months (EORTC QLQ C30) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 months (EORTC QLQ C30) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 weeks (EORTC QLQ BN20) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 3 months (EORTC QLQ BN20) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 months (EORTC QLQ BN20) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 weeks (EQ-5D) | 6 weeks postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 3 months (EQ-5D) | 3 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 6 months (EQ-5D) | 6 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Serious Adverse Events | 6 weeks postoperatively
  Serious Adverse Events within 6 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Gerritsen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Hospital Leuven, Leuven, Belgium
- Germany (2):
  - University Hospital Heidelberg, Heidelberg
  - Technical University Munich, Munich
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Medical Center Haaglanden, The Hague, South Holland
- Inselspital Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided